CLINICAL TRIAL: NCT07322445
Title: Development and Identification of Magnetic Resonance, Electrophysiological, and Fiber-optic Imaging Biomarkers of Myofascial Pain
Brief Title: Multi-modal Imaging of Myofascial Pain - Phase 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Yong Wang, Principal Investigator, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202506118; R33AT012283 (NIH)
Record Dates: First submitted 2025-10-06; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Myofascial Pain
Keywords: Magnetic Resonance Imaging; Surface Electromyography; Fiber-optic Imaging and Sensing
MeSH Terms: interventions — Injections; Bupivacaine; Dry Needling

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemical Injection (Active Comparator): Local chemical injection at clinician-identified myofascial trigger points.
  Interventions: Drug: 50/50 Mixture of Lidocaine 1% injection + Bupivacaine 0.25% Injectable Solution
- Dry Needle (Placebo Comparator): Dry needling at clinician-identified myofascial trigger points.
  Interventions: Procedure: Dry Needling

INTERVENTIONS:
Drug: 50/50 Mixture of Lidocaine 1% injection + Bupivacaine 0.25% Injectable Solution — Treatment Group: Receives trigger-point injection with a 50/50 mixture of 1% lidocaine and 0.25% bupivacaine
  Arms: Chemical Injection
Procedure: Dry Needling — Single session of dry needling to the identified trigger point(s) per protocol.
  Arms: Dry Needle

SUMMARY:
The goal of this study is to evaluate imaging biomarkers for quantitative assessments of myofascial pain and determine their ability to monitor treatment response and predict clinical outcomes.

DETAILED DESCRIPTION:
This Phase 2 randomized clinical trial builds upon findings from Phase 1, which identified candidate imaging biomarkers of myofascial pain. The study will assess whether these biomarkers can monitor responses to local chemical injection treatment and predict clinical outcomes.

Participants with neck/shoulder pain and the presence of active myofascial trigger points will be referred from pain management clinics or recruited through the Volunteer for Health office. Eligible participants will undergo multi-modal imaging procedures, including magnetic resonance imaging (MRI), surface electromyography (sEMG), and fiber-optic imaging. Participants will then be randomized to receive either chemical injection or dry needling at the identified trigger points.

Over the course of two study visits, spaced approximately two weeks apart, participants will complete imaging procedures and patient-reported outcome questionnaires. The study team will analyze imaging and clinical data to evaluate the capacity of identified biomarkers to detect treatment-related changes and to predict longer-term clinical response.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between the ages of 18 and 80 years old.
2. History of spontaneous (non-provoked) pain in the neck and/or shoulder region lasting at least 3 months. Neck and/or shoulder pain, unilateral or bilateral.
3. Presence of a palpable myofascial trigger point (MTrP) in one or both upper trapezius muscles.
4. The participant has a Numeric Pain Rating Scale of 4/10 or more in the last one week, and the pain is reproducible by palpating the trigger point.
5. Pain localized to the area of the trigger point that is reproduced or worsened upon palpation.
6. Radiation of pain to the head, neck, or face with palpation is allowed but not required.

Exclusion Criteria:

1. Age <18 or >80 years old.
2. Acute cervical spine pathology, trauma (e.g. whiplash) or cervical radiculopathy
3. History of surgery involving the head, neck, or shoulder girdle.
4. Presence of neuromuscular pathologies or inflammatory muscle diseases (e.g. dermatomyositis)
5. Systemic disease with diffuse body pain (e.g. system lupus erythematosus)
6. Peripheral neuropathy
7. Cancer-related pain
8. Pregnancy, coagulopathy or other bleeding disorder, fever, general/local infection at the pain site, substance abuse, or any other diseases that may account for signs and symptoms mimicking myofascial pain.
9. Contraindication to MRI
10. Chronic fatigue syndrome, fibromyalgia, or chronic Lyme disease.
11. Use of acupuncture or changes in pain medications within 6 weeks of enrollment.
12. Receipt of Botox injection to the neck/shoulder region within the past 3 months or trigger point injection within the past 6 weeks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Statistical Plan | Baseline and follow-up study visits approximately 2 weeks apart (each visit lasting 3-4 hours)
  The statistical analysis will assess the ability of imaging biomarkers to distinguish pathological and physiological differences among participant groups. Imaging biomarkers of the myofascial tissue will be measured for each participant, including tissue stiffness, hydration, inflammation, blood oxygenation and flow, and electrical activity. Group differences in each imaging biomarker will be evaluated independently using Student's t-test or Wilcoxon rank-sum test, as appropriate. Each biomarker will be analyzed and reported separately and will not be combined into a composite measure. We hypothesize that some imaging biomarkers will demonstrate large effect sizes between participant groups. Statistical power will be estimated based on Cohen's d for individual biomarkers. With an expected effect size greater than 0.9, the proposed sample size provides greater than 80% power. Multi-modal imaging is expected to identify biomarkers with strong group differences.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No